CLINICAL TRIAL: NCT01448486
Title: A Randomised Controlled Clinical Trial of the Efficacy of HAART Intensification With Raltegravir in HIV Virally Suppressed Patients With Cognitive Impairment
Brief Title: A Study of the Neurological Effects of Adding Raltegravir to HAART Regimen in Patients With HIV
Acronym: HANDral
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding withdrawn based on unacceptably slow recruitment rate.
Sponsor: St Vincent's Hospital, Sydney (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Bruce Brew, Professor, St Vincent's Hospital, Sydney
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/033; IISP 37693 (Other Grant/Funding Number: Merck Sharp & Dohme)
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Results first posted 2014-01-03 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-05

CONDITIONS: Human Immunodeficiency Virus (HIV); HIV Associated Neurocognitive Disorders (HAND)
Keywords: HIV; HAND; Human Immunodeficiency Virus; Raltegravir; HIV Associated Neurocognitive Disorders; Neuro-HAART; Neurocognitive; Neurology
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care HAART (No Intervention): Participants randomised to this arm will remain on their standard of care Highly Active Antiretroviral Therapy (HAART).
- Raltegravir (Experimental): Participants randomised to this arm will remain on their standard of care Highly Active Antiretroviral Therapy (HAART) with the addition of Raltegravir 400 mg twice daily (BID).
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Oral raltegravir, 400 mg tablet, twice daily for one year.
  Other Names: Isentress
  Arms: Raltegravir

SUMMARY:
HIV related cognitive impairment still occurs despite highly active antiretroviral therapy (HAART). HIV disease affects the brain in 20-40% of patients with advancing HIV disease leading to varying degrees of cognitive impairment, recently termed HIV associated neurocognitive disorders (HAND).

HAND may occur in patients who are virally suppressed in both blood and CSF. Patients with HIV Associated Neurological Disorders (HAND) who are virally suppressed in both their blood and cerebrospinal fluid (CSF), whilst on a highly active antiretroviral therapy (HAART) regimen may have significant cognitive improvement with HAART intensification with the medication Raltegravir; compared to those who remain on their existing regimen.

This study will be a prospective, interventional, randomised and unblinded controlled clinical trial. The aim of this study will be to determine whether HAART intensification with the medication Raltegravir, leads to significant improvement in HIV associated neurological disorders (HAND).

Patients with the recent progression (within 6 months) of HAND (validated by neuropsychological assessment) on HAART who are virally suppressed (<50 copies per ml) in blood and CSF will be randomised to have their existing HAART regimen intensified with raltegravir 400mg twice daily, or not. The control arm will remain on their medication regimen as prescribed. The target is to enrol 110 patients into the control group, and 110 patients into the Raltegravir intensification group.

Patients will undergo baseline neuropsychological testing, MRI, blood tests, and cerebral spinal fluid (CSF) tests (via a lumbar puncture). The methods used to determine the effectiveness of adding Raltegravir, will include further neuropsychological testing at 6 months; and neuropsychological testing, MRI and CSF assessment at 12 months. Neuropsychological testing completed at 6 and 12 months will be completed by a "blind assessor", in that they will have no knowledge of which arm (treatment or control) the participant is enrolled in.

An evaluation (neuropsychological testing) will be performed should the patient deteriorate during the course of the study, as recognised by the patient's managing physician. The decision of the Antiretroviral medication regimen to be used in such a case will be determined by the managing physician. At the end of the study protocol (12 months) the patient's HAART therapy will be managed by their primary physician.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* On HAART, with plasma HIV viral load < 50 copies/ml for previous 12 months or more
* Able to provide informed consent
* HAND diagnosis, with symptom progression within previous 6 months (while on existing HAART regimen)

Exclusion Criteria:

* Non-HIV related neurological disorders and active CNS opportunistic infection (as assessed by full blood count, electrolytes, creatinine, glucose, LFT's, cryptococcal antigen, VDRL, MRI brain scan and CSF fluid analysis for cell count, protein, glucose, culture, VDRL and cryptococcal antigen)
* Psychiatric disorders on the psychotic axis
* Current major depression
* Current substance use disorder, or severe substance use disorders within 12 months of study entry
* Active HCV (detectable HCV RNA)
* History of loss of consciousness > 1 hour
* Non-proficient in English
* Medications known to pharmacologically interact with ARV's
* Currently taking an Integrase Inhibitor
* Pregnancy (as assessed by the urine pregnancy test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J Brew, MBBS, PhD, Principal Investigator — St Vincent's Hospital, Sydney
Locations (2):
- Australia (2):
  - St. Vincent's Hospital, Sydney, New South Wales
  - The Alfred Hospital, Melbourne, Victoria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from October 2011 to October 2013. Participants were known patients of the PI or referred from local tertiary sexual health clinics by associate investigators.
Groups:
- Raltegravir: Participants randomised to this arm will remain on their standard of care Highly Active Antiretroviral Therapy (HAART) with the addition of Raltegravir 400 mg twice daily (BID).
  Raltegravir : Oral raltegravir, 400 mg tablet, twice daily for one year.
Period: Overall Study
Arm/Group | Raltegravir | Standard of Care HAART
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir | Standard of Care HAART | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (8.7) | 59.3 (4.9) | 55.7 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Neurocognitive Function
Description: Change in overall neurocognitive performance, defined as a global neurocognitive z-score, over the study time-period (baseline, 6-months, 12-months). To derive this score, 1) raw scores obtained from a 5-domain brief neurocognitive battery were converted to age-corrected z-scores (M=0, SD=1) and 2) the set of individual subtest z-scores were averaged to generate a single composite (global) z-score for each subject. Lower (negative) scores therefore indicate greater levels of cognitive impairment.
Time Frame: Baseline, 6 months and 12 months
Population: Study was terminated prematurely with an incomplete study dataset any before any meaningful statistical analysis of the data (including change over the study time-points) could be performed.
Measure: Mean (Standard Error); unit: Global Neurocognitive Z-Score
Arm/Group | Raltegravir | Standard of Care HAART
Number analyzed (Participants) | 3 | 3
Global Neurocognitive Z-Score
  Baseline | -0.83 (0.29) | -0.39 (0.20)
  6 months | -0.55 (0.12) | -0.48 (0.45)
  12 months | -0.47 (0.46) | -0.54 (0.32)

2. Secondary Outcome: Cerebrospinal Fluid
Description: To determine if there is improvement in CSF neopterin concentrations with the addition of Raltegravir.
Time Frame: Baseline and 12 months
Population: Study was terminated prematurely with an incomplete study dataset before any meaningful analyses of the data could be conducted. CSF was not collected at 12 months for n=1 raltegravir and n=1 control who refused lumbar puncture.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Raltegravir | Standard of Care HAART
Number analyzed (Participants) | 3 | 3
nmol/L
  Baseline | 11.67 (2.91) | 34.00 (16.26)
  12 months | 17.00 (7.00) | 12.00 (3.00)

ADVERSE EVENTS:
Arm/Group | Raltegravir | Standard of Care HAART
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir (N=3) | Standard of Care HAART (N=3)
Muscle strain (General disorders) | 1 (1) | 0
Flu-like illness (General disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to incomplete dataset with sample size too small to produce any meaningful statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No